CLINICAL TRIAL: NCT04272801
Title: Pre-Operative Window of Adjuvant Endocrine Therapy to Inform Radiation Therapy Decisions In Older Women With Early-Stage Breast Cancer
Brief Title: Pre-Operative Window of Adjuvant Endocrine Therapy to Inform RT Decisions in Older Women With Early-Stage Breast Cancer
Acronym: POWER
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shayna Showalter, MD (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor-Investigator, Shayna Showalter, MD, Sponsor-Investigator, University of Virginia
Organization: University of Virginia (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 22040; 5R21CA277311-02 (NIH)
Record Dates: First submitted 2020-02-04; First posted 2020-02-17 (Actual); Results first posted 2025-10-22 (Actual); Last update posted 2025-10-22 (Actual); Status verified 2025-09

CONDITIONS: Breast Cancer Female
Keywords: breast cancer; endocrine therapy; radiation; letrozole; anastrozole; exemestane; tamoxifen; survey; questionnaire; geriatric
MeSH Terms: conditions — Breast Neoplasms | interventions — Tamoxifen; Letrozole; Anastrozole; exemestane; Patient Reported Outcome Measures; Surveys and Questionnaires

STUDY DESIGN:
Intervention Model Description: Pilot, 1 arm
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Pre-operative endocrine therapy (Experimental): All participants enrolled to the study will receive 3 months of pre-operative endocrine therapy (e.g. tamoxifen or aromatase inhibitors (AIs) such as letrozole, anastrozole, or exemestane). The choice and dose of endocrine therapy will be at the discretion of the treating medical oncologist.
  Interventions: Drug: tamoxifen, letrozole, anastrozole, or exemestane; Behavioral: Patient reported outcomes

INTERVENTIONS:
Drug: tamoxifen, letrozole, anastrozole, or exemestane — choice and dose of neoadjuvant endocrine therapy at the discretion of the treating medical oncologist
  Other Names: Endocrine therapy
Behavioral: Patient reported outcomes — Questionnaire inquiries include the following:
  * how cancer affects daily living
  * beliefs about medicines and sensitivity to medicine
  * symptoms
  * adherence to endocrine therapy
  * general health and well being
  * depression and anxiety
  * preference regarding radiation therapy
  Other Names: surveys, questionnaires

SUMMARY:
This is a prospective multisite exploratory study for women ≥ 65 years of age with early stage estrogen receptor positive (ER+) breast cancer. These individuals will be treated with 3 months of pre-operative endocrine therapy (pre-ET) with assessment of tolerance to the endocrine therapy by patient reported outcome (PRO) measures (patient surveys).

DETAILED DESCRIPTION:
This single arm pilot study evaluates the use of pre-operative endocrine therapy in women with early stage ER+ breast cancer who are 65 years or older and are scheduled to have breast conservation surgery (BCS). The purpose of this study is to see if tolerance of pre-operative endocrine therapy helps inform decisions on whether or not to omit radiation. Participants will be treated with the novel approach of 3 months of pre-operative endocrine therapy, so that the participants and providers will have some indication of tolerance prior to making a decision about radiation omission. Tolerance of the endocrine therapy will be assessed by patient reported outcome (PRO) measures during neoadjuvant and adjuvant endocrine therapy treatment periods. Breast cancer participants and their surgical oncologists will be asked their preference regarding radiation therapy before starting endocrine therapy and again pre-operatively. They will make a determination regarding radiation therapy as per standard care. The hypothesis is that knowledge of tolerance of endocrine therapy will influence the decision by the patient and the surgical oncologist whether or not to elect radiation omission.

ELIGIBILITY:
Inclusion Criteria (Summary):

* ECOG performance status 0-2
* Diagnosed with anatomic stage I, ER positive, PR positive or negative, and HER2 non amplified invasive breast cancer and clinically negative nodes; any invasive breast cancer histologic subtype may be enrolled
* Tumor size ≤ 2 cm
* Patient has elected BCS as surgical choice
* Eligible to receive tamoxifen or an aromatase inhibitor
* Ability to take oral medication and be willing to adhere to the endocrine therapy for the 3 month period prior to BCS

Exclusion Criteria (Summary):

* Prior or current use of endocrine therapy for breast cancer
* History of ipsilateral breast radiation
* Pregnancy or lactation
* Has a known additional malignancy that is progressing or requires active treatment. Exceptions include basal cell carcinoma of the skin or squamous cell carcinoma of the skin that has undergone potentially curative therapy or in situ cervical cancer.
* Current or planned use of a strong CYP2D6 inhibitor (e.g. Fluoxetine, Paroxetine) and is not able to receive an endocrine therapy agent that does not use the CYP2D6 pathway

Min Age: 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 84 (Actual)
Dates: Start 2020-04-07 (Actual); Primary Completion 2024-06-05 (Actual); Study Completion 2026-06-01 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Shayna L Showalter, MD, Principal Investigator — University of Virginia
Locations (2):
- United States (2):
  - University of Virginia, Charlottesville, Virginia
  - Virginia Commonwealth University Massey Cancer Center, Richmond, Virginia

RESULTS

PARTICIPANT FLOW:
Groups:
- Pre-operative endocrine therapy: All participants enrolled to the study will receive 3 months of pre-operative endocrine therapy (e.g. tamoxifen or aromatase inhibitors (AIs) such as letrozole, anastrozole, or exemestane). The choice and dose of endocrine therapy will be at the discretion of the treating medical oncologist.
  tamoxifen, letrozole, anastrozole, or exemestane: choice and dose of neoadjuvant endocrine therapy at the discretion of the treating medical oncologist
  Patient reported outcomes: Questionnaire inquiries include the following:
  * how cancer affects daily living
  * beliefs about medicines and sensitivity to medicine
  * symptoms
  * adherence to endocrine therapy
  * general health and well being
  * depression and anxiety
  * preference regarding radiation therapy
Period: Overall Study
Arm/Group | Pre-operative endocrine therapy
Started | 84
Completed | 75
Not Completed | 9
Not completed — Withdrawal by Subject | 4
Not completed — Lost to Follow-up | 4
Not completed — Ineligible | 1

BASELINE CHARACTERISTICS:
Population: A total of 84 participants consented. One was found ineligible after consent, leaving 83 as the baseline. Of these, 4 withdrew and 4 were lost to follow-up. Data from 75 participants were analyzed for baseline characteristics.
Arm/Group | Pre-operative endocrine therapy
Number analyzed (Participants) | 75
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 0
  >=65 years | 75
Age, Continuous [Median (Full Range); unit: years] | 78.5 [65 to 92]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 75
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 74
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 7
  White | 68
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 75

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Changed Their Preference for Adjuvant Radiation Treatment
Description: Change in participant response to question regarding preference for adjuvant radiation treatment
Time Frame: up to 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Pre-operative endocrine therapy
Number analyzed (Participants) | 75
Participants | 21

2. Primary Outcome: Change in Surgeon Preference for Adjuvant Radiation Treatment
Description: Change in surgical oncologist response to question regarding preference for adjuvant radiation treatment
Time Frame: up to 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Pre-operative endocrine therapy
Number analyzed (Participants) | 75
Participants | 18

3. Secondary Outcome: Health Related Quality of Life Surveys as Predictive Measure for Endocrine Therapy Adherence and to Assess Effect of Pre-ET on Decision Outcomes for Adjuvant Therapy After BCS
Description: Health related quality of life will be assessed using the EORTC QLQ-C30 and QLQ-BR23.
Time Frame: Through 24 months after start of adjuvant treatment period
Reporting Status: Not Posted

4. Secondary Outcome: General Symptom Burden as Predictive Measure for Endocrine Therapy Adherence and to Assess Effect of Pre-ET on Decision Outcomes for Adjuvant Therapy After BCS
Description: General symptom burden will be assessed using the Breast Cancer Prevention Trial Symptom Checklist.
Time Frame: Through 24 months after start of adjuvant treatment period
Reporting Status: Not Posted

5. Secondary Outcome: Illness Perception as Predictive Measure for Endocrine Therapy Adherence and to Assess Effect of Pre-ET on Decision Outcomes for Adjuvant Therapy After BCS
Description: Illness perception will be assessed using the Brief Illness Perception Questionnaire.
Time Frame: Through 24 months after start of adjuvant treatment period
Reporting Status: Not Posted

6. Secondary Outcome: Beliefs About Medicine as Predictive Measure for Endocrine Therapy Adherence and to Assess Effect of Pre-ET on Decision Outcomes for Adjuvant Therapy After BCS
Description: Beliefs about medicine will be assessed using the Beliefs about Medicines Questionnaire.
Time Frame: Through 24 months after start of adjuvant treatment period
Reporting Status: Not Posted

7. Secondary Outcome: Perceived Sensitivity to Medicine as Predictive Measure for Endocrine Therapy Adherence and to Assess Effect of Pre-ET on Decision Outcomes for Adjuvant Therapy After BCS
Description: Perceived sensitivity to medicine will be assessed using the Perceived Sensitivity to Medicine Scale.
Time Frame: Through 24 months after start of adjuvant treatment period
Reporting Status: Not Posted

8. Secondary Outcome: Breast Cancer Beliefs as Predictive Measure for Endocrine Therapy Adherence and to Assess Effect of Pre-ET on Decision Outcomes for Adjuvant Therapy After BCS
Description: Breast cancer beliefs will be assessed using the UVA Breast Cancer Belief Survey, a novel series of questions regarding patient beliefs about breast cancer and breast cancer medications.
Time Frame: Through 24 months after start of adjuvant treatment period
Reporting Status: Not Posted

9. Secondary Outcome: Treatment Decision as Predictive Measure for Endocrine Therapy Adherence and to Assess Effect of Pre-ET on Decision Outcomes for Adjuvant Therapy After BCS.
Description: Treatment decision will be assessed using the Treatment Decision Survey, a novel series of questions regarding why subjects decide to have or not to have radiation therapy, and why or why not to restart endocrine therapy.
Time Frame: up to 90 days after surgery, chemotherapy completion, or RT completion, whichever is later
Reporting Status: Not Posted

10. Secondary Outcome: Perceptions Related to Medical Choices as Predictive Measure for Endocrine Therapy Adherence and to Assess Effect of Pre-ET on Decision Outcomes for Adjuvant Therapy After BCS.
Description: Subjects' perceptions related to their medical choices will be assessed using the Decisional Conflict Scale and the Decision Regret Scale.
Time Frame: Through 24 months after start of adjuvant treatment period
Reporting Status: Not Posted

11. Secondary Outcome: Depression and Anxiety as Predictive Measure for Endocrine Therapy Adherence
Description: Depression and anxiety will be assessed using the Center for Epidemiologic Studies Depression Scale Revised.
Time Frame: Through 24 months after start of adjuvant treatment period
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the date of informed consent through 30 days after the last dose of neo-adjuvant endocrine therapy for non-serious AEs, and through study completion (an average of approximately 27 months) for related SAEs or until initiation of another therapy.
Arm/Group | Pre-operative endocrine therapy
All-Cause Mortality (participants affected / at risk) | 0/75
Serious Adverse Events (participants affected / at risk) | 2/75
Other Adverse Events (participants affected / at risk) | 35/75
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pre-operative endocrine therapy (N=75)
Pulmonary Embolism (Vascular disorders) | 1 (1)
Acute Stroke (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pre-operative endocrine therapy (N=75)
Agitation (Psychiatric disorders) | 1 (1)
Alanine aminotransferase (ALT) Increase (Investigations) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 9 (9)
Anxiety (Psychiatric disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 13 (13)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Aspartate aminotransferase (AST) Increase (Investigations) | 1 (1)
Back Pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Bladder Infection (Infections and infestations) | 2 (3)
Blurred Vision (Eye disorders) | 2 (2)
Constipation (Gastrointestinal disorders) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 3 (3)
Dizziness (Nervous system disorders) | 1 (1)
Dry Mouth (Gastrointestinal disorders) | 1 (1)
Dry Skin (Skin and subcutaneous tissue disorders) | 2 (2)
Edema Limbs (General disorders) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 2 (2)
Fatigue (General disorders) | 13 (14)
Fever (General disorders) | 1 (1)
Flank Pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Flu Like Symptoms (General disorders) | 1 (1)
Covid-19 (General disorders) | 1 (1)
Insomnia (Psychiatric disorders) | 7 (7)
Headaches (Nervous system disorders) | 6 (6)
Hot Flashes (Vascular disorders) | 22 (22)
Hypercalcemia (Metabolism and nutrition disorders) | 1 (1)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (1)
Hypertension (Vascular disorders) | 3 (3)
Hyperglycemia (Investigations) | 1 (1)
Joint Effusion (Musculoskeletal and connective tissue disorders) | 1 (1)
Lung Infection (Infections and infestations) | 1 (1)
Lymphocyte Count Increased (Investigations) | 1 (1)
Memory Impairment (Nervous system disorders) | 1 (1)
Vitamin D Deficiency (Metabolism and nutrition disorders) | 1 (1)
Mucositis Oral (Gastrointestinal disorders) | 1 (1)
Muscle Cramp (Musculoskeletal and connective tissue disorders) | 2 (2)
Neck/Bilateral Arm Pressure (Musculoskeletal and connective tissue disorders) | 1 (1)
Knee Pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Transient Joint Stiffness (Musculoskeletal and connective tissue disorders) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2)
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 5 (5)
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
Perineal Pain (Reproductive system and breast disorders) | 1 (1)
Pruritis (Skin and subcutaneous tissue disorders) | 2 (2)
Mood Swings (Psychiatric disorders) | 1 (1)
Rash Maculo-Papulr (Skin and subcutaneous tissue disorders) | 1 (1)
Thromboembolic Event (Vascular disorders) | 1 (2)
Transient Ischemic Attacks (Nervous system disorders) | 1 (1)
Upper Respiratory Infection (Infections and infestations) | 1 (1)
Urinary Incontinence (Renal and urinary disorders) | 1 (1)
Urinary Tract Infection (Infections and infestations) | 1 (1)
Uterine Pain (Reproductive system and breast disorders) | 1 (1)
Vagina Dryness (Reproductive system and breast disorders) | 2 (2)
Vaginal Infection (Infections and infestations) | 1 (1)
Vaginal Pain (Reproductive system and breast disorders) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 1 (1)
Vision Decrease (Eye disorders) | 1 (1)
Weight Loss (Investigations) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-02-21): https://cdn.clinicaltrials.gov/large-docs/01/NCT04272801/Prot_SAP_000.pdf
  • Informed Consent Form (2023-01-10): https://cdn.clinicaltrials.gov/large-docs/01/NCT04272801/ICF_001.pdf